CLINICAL TRIAL: NCT07299617
Title: The Effect of Lavender Oil Applied Via Inhalation On Headache And Anxiety Level in Individuals Undergoing Hemodialysis Treatment
Brief Title: The Effect of Lavender Oil Applied Via Inhalation on Headache and Anxiety Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Goknur Demir Hacimusalar (Other)
Responsible Party: Sponsor-Investigator, Goknur Demir Hacimusalar, Phd, TC Erciyes University
Organization: TC Erciyes University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ERU-SBF-GDH-01
Record Dates: First submitted 2025-09-22; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Hemodialysis Patients
Keywords: Hemodialysis; Pain; Anxiety; Lavender oil; Nursing
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Aromatherapy; lavender oil

STUDY DESIGN:
Intervention Model Description: It was conducted as a randomized controlled study to determine the effect of pure lavender oil applied by inhalation for 5 minutes, 3 times a week, for a month, on the severity of headaches that develop during dialysis and the level of state-trait anxiety in individuals receiving hemodialysis treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pure Lavender Oil Inhalation Group (Other): Participants assigned to the lavender oil inhalation intervention.
  Interventions: Other: Lavender Oil Inhalation
- Control group patients. (Other): A total of 32 control group patients (standard hemodialysis care)
  Interventions: Other: Standard Hemodialysis Care

INTERVENTIONS:
Other: Lavender Oil Inhalation — Participants receive pure medical lavender oil (Lavandula angustifolia) with a certificate of analysis. During the 2nd hour of the dialysis session, 3 drops of lavender oil are applied to a 6x6 cm gauze pad. Patients are instructed to inhale the scent from a distance of 5 cm for 5 minutes. This procedure is performed 3 times a week for 4 weeks, totaling 12 sessions. The dosage adjustment and application are performed by the researchers.
  Other Names: Aromatherapy with Lavender Oil; Lavandula angustifolia inhalation
  Arms: Pure Lavender Oil Inhalation Group
Other: Standard Hemodialysis Care — Participants in the control group receive only routine hemodialysis treatment. No additional aromatherapeutic intervention or inhalation is administered during the study period.
  Arms: Control group patients.

SUMMARY:
This randomized controlled study aims to determine the effect of pure lavender oil inhalation on headache severity and anxiety levels in hemodialysis (HD) patients. The research, conducted in three dialysis centers, included a total of 62 patients who were randomly assigned to either an intervention group (n=30) receiving lavender oil inhalation or a control group (n=32) receiving standard care. Data were collected using the Visual Analogue Scale (VAS) for headache severity and the State-Trait Anxiety Inventory (STAI) for anxiety levels.

DETAILED DESCRIPTION:
Background: Pain, particularly headaches, is a common symptom in hemodialysis (HD) patients that can significantly impact their quality of life. This study investigates the potential therapeutic effect of an integrative medicine approach-lavender oil inhalation-as a non-pharmacological intervention.

Study Design: This is a multi-center, prospective, randomized, open-label, parallel-assignment controlled study. The study population consists of 62 adult hemodialysis patients from three dialysis centers in a city center in Turkey. Participants were enrolled based on specific inclusion criteria, including experiencing headaches during HD sessions.

Interventions: Patients were randomly assigned to one of two groups. The intervention group (n=30) received pure lavender oil inhalation for 5 minutes, three times a week, at the 2nd hour of their HD session, for a duration of one month. The control group (n=32) continued to receive only their standard hemodialysis care without any additional intervention.

Data Collection and Outcome Measures: Data were collected using a patient introduction form to gather demographic information. For a period of four weeks, headache severity was measured using the Visual Analogue Scale (VAS) immediately before, two hours after the start, and at the end of each dialysis session. Anxiety levels were assessed using the State-Trait Anxiety Inventory (STAI), with the STAI-S applied at the 2nd and 4th hours of dialysis and the STAI-T at the beginning and end of the four-week study period.

ELIGIBILITY:
Inclusion Criteria:

* Those who are 18 years of age and over,

  * Able to understand and communicate in Turkish,
  * Receiving hemodialysis treatment three times a week for at least 3 months,
  * Not pregnant and not planning a pregnancy,
  * Having a pain intensity of 3 or more on the Visual Analog Scale, measured twice,
  * Headache that develops during dialysis,
  * Headache worsening throughout the dialysis session,
  * Headache resolves spontaneously within 72 hours after dialysis ends,
  * No visual or hearing impairment,
  * Individuals who could take painkillers when they had pain were included in the study

Exclusion Criteria:

* Those who are allergic to or uncomfortable with the smell of lavender oil,

  * Having any obstacle to smell,
  * Having a history of asthma,
  * Individuals who used other complementary integrative medicine methods during the treatment process were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Headache Severity measured by Visual Analog Scale (VAS). | Measured 3 times during each hemodialysis session (immediately before, 2 hours after start, and at the end of dialysis) over a period of 4 weeks (total of 12 sessions).
  Headache severity is measured using a 10-unit Visual Analog Scale (VAS) where "0" represents no pain and "10" represents the most severe pain possible. A lower score indicates a reduction in headache intensity

SECONDARY OUTCOMES:
State Anxiety Levels measured by State Anxiety Inventory (STAI-S). | Measured at the 2nd and 4th hours of dialysis sessions throughout the 4-week study period.
  This inventory consists of 20 items measuring how the individual feels at a given moment. Scores range from 20 to 80, with higher scores indicating higher levels of anxiety.
Trait Anxiety Level (STAI-T) | At the beginning of the study (baseline) and at the end of the 4th week.
  Measured by the State-Trait Anxiety Inventory - Trait subscale (20 items). Scores range from 20 to 80, where higher scores indicate higher general levels of anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes Univercity, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data (IPD) will be shared. Supporting documents such as the study protocol and clinical study report will also be available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 6 months after publication of the study results, and will be available for 10 years.
Access Criteria: The data will be available upon request by contacting the corresponding author via email. The requester must sign a data access agreement.